CLINICAL TRIAL: NCT05987514
Title: Role of Dynamic Contrast-Enhanced Ultrasound (D-CEUS) and Shear-wave Elastography (SWE) in Predicting Response to Locoregional Treatments and Disease Recurrence in Patients Affected by Hepatocellular Carcinoma (HCC)
Brief Title: Multimodal Ultrasound and Hepatocellular Response to Local Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4175
Record Dates: First submitted 2023-03-16; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients affected by hepatocellular carcinoma needing to undergo loco-regional treatment
  Interventions: Diagnostic Test: multimodal ultrasound

INTERVENTIONS:
Diagnostic Test: multimodal ultrasound — contrast-enhanced ultrasound and shear wave elastography on liver target lesion

SUMMARY:
Consecutive patients with HCC who should undergo to locoregional treatments (ablation or trans-arterial chemoembolization) according to international guidelines will be enrolled. atients will undergo CEUS and SWE before and after 24 hours from the procedure as per clinical practice in our center. Subsequently, the patients will continue the normal follow-up which includes control computed tomography/magnetic resonance one month after treatment and subsequently every three months.

DETAILED DESCRIPTION:
Primary objective: To evaluate the correlation between pre-treatment ultrasound parameters (D-CEUS and elastography) and one-month response to therapy evaluated with contrast-enhanced computed tomography.

Secondary objective: To identify quantitative ultrasound parameters able to predict overall survival and disease-free survival.

Study design: Prospective single-center study. Methods: 50 consecutive patients with HCC who should undergo to locoregional treatments (ablation or trans-arterial chemoembolization) according to international guidelines will be enrolled in the Unit of Internal Medicine and Gastroenterology of the Policlinico Gemelli. After obtaining informed consent and identifying the target lesion in B-mode ultrasound, patients will undergo CEUS and SWE before and after 24 hours from the procedure as per clinical practice in our center. Subsequently, the patients will continue the normal follow-up which includes control computed tomography/magnetic resonance one month after treatment and subsequently every three months. In addition, the personal, clinical and laboratory data necessary to determine the hepatological scores of disease severity such as MELD and Child-Pugh will be collected. The study has an expected duration of one year.

ELIGIBILITY:
Inclusion Criteria adult patients with single nodule hepatocellular carcinoma detectable with B-mode ultrasound and scheduled for locoregional treatment

Exclusion Criteria:

* liver failure
* previous treatments fo hepatocellular carcinoma
* chronic or acute heart failure
* known ipersesitivity to ultrasound contrast agent
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
predicting HCC response to treatment | one month after local treatment
  to quantify peak enhancement intensity in Arbitray Units AU(measured by analysing D-CEUS time-intensity curves) in patients undergoing local treatments for HCC, stratified according to one-month treatment response (responders or non-responders) assessed by computed tomography

SECONDARY OUTCOMES:
predicting HCC response to treatment | one month after local treatment
  to quantify mean HCC stiffness in patients undergoing local treatments for HCC, stratified according to one-month treatment response (responders or non-responders) assessed by computed tomography
predicting overall survival | 12 months after treatment
  to identify association between the peak enhancement intensity in Arbitray Units AU (measured by analysing D-CEUS time-intensity curves) in patients undergoing local treatments for HCC and time of survival
predicting disease-free survival | 12 months after treatment
  to identify the association between the peak enhancement intensity in Arbitray Units AU (measured by analysing D-CEUS time-intensity curves) in patients undergoing local treatments for HCC and time of disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy